CLINICAL TRIAL: NCT05342467
Title: Gemeprost Versus Dinoprostone in the Medical Management of First Trimester Miscarriages: a Randomized Controlled Study
Brief Title: Gemeprost Versus Dinoprostone in First Trimester Miscarriages
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF-2021-504
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Missed Abortion; Medical; Abortion, Fetus; Incomplete Abortion
Keywords: miscarriages; first trimester; medical treatment
MeSH Terms: conditions — Abortion, Missed; Abortion, Incomplete; Abortion, Spontaneous | interventions — gemeprost; Suppositories; Dinoprostone

STUDY DESIGN:
Intervention Model Description: Comparison between intravaginal gemeprost and dinoprostone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemeprost (Active Comparator): Gemeprost 1 mg inserted 3 hourly for maximum of 5 doses in 24 hours.
  Interventions: Drug: Gemeprost 1 Mg Vaginal Pessary; Drug: Dinoprostone 3 mg
- Dinoprostone (Active Comparator): Dinoprostone 3 mg inserted 4 hourly for maximum of 3 doses in 24 hours.
  Interventions: Drug: Gemeprost 1 Mg Vaginal Pessary; Drug: Dinoprostone 3 mg

INTERVENTIONS:
Drug: Gemeprost 1 Mg Vaginal Pessary — Intravaginal gemeprost 1 mg inserted 3 hourly for maximum of 5 doses in 24 hours
Drug: Dinoprostone 3 mg — Intravaginal dinoprostone 3 mg inserted 4 hourly for maximum of 3 doses in 24 hours

SUMMARY:
Comparison between gemeprost and dinoprostone to evacuate first trimester miscarriages.

DETAILED DESCRIPTION:
Women who are diagnosed with first trimester missed miscarriages are invited to participate in the study. They will be randomised to either gemeprost or dinoprostone.

ELIGIBILITY:
Inclusion Criteria:

* missed miscarriages
* incomplete miscarriages
* first trimester

Exclusion Criteria:

* coagulopathy
* Rhesus negative
* suspected ectopic pregnancy or pregnancy of unknown location
* on anticoagulation drug
* septic miscarriages
* hemodynamically unstable

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Percentage of women who achieved complete evacuation | from recruitment until up to one week after commencement of treatment
  Complete expulsion of product of conception

SECONDARY OUTCOMES:
Percentage of women who experienced side effects | from recruitment until up to one week after commencement of treatment
  side effects towards each drug such as fever, gastrointestinal upset

CONTACTS AND LOCATIONS:
Overall Officials: Rahana Abd Rahman, Principal Investigator — National University of Malaysia
Locations (2):
- Malaysia (2):
  - UKM Medical Center, Kuala Lumpur, W.Persekutuan
  - UKM Medical Centre, Kuala Lumpur, W.Persekutuan

IPD SHARING:
Plan to Share IPD: Undecided
Yes